CLINICAL TRIAL: NCT05111366
Title: An Open, Single Arm, Multicenter, Exploratory Phase II Clinical Trial of TQB2450 Plus Anlotinib as Adjuvant Therapy in HCC Patients at High Risk of Recurrence After Resection
Brief Title: TQB2450 Plus Anlotinib as Adjuvant Therapy in HCC Patients at High Risk of Recurrence After Resection
Acronym: ALTER-H006
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xianhai Mao (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Xianhai Mao, Professor, Hunan Provincial People's Hospital
Organization: Hunan Provincial People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210727
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Hepatocellular Carcinoma; Adjuvant Therapy
Keywords: HCC; Adjuvant Therapy; TQB2450; Anlotinib
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2450 injection combined with Anlotinib hydrochloride capsules (Experimental)
  Interventions: Drug: TQB2450 injection; Drug: Anlotinib hydrochloride capsules

INTERVENTIONS:
Drug: TQB2450 injection — TQB2450 is an injection in the form of 1200mg, ivgtt, q3W.
Drug: Anlotinib hydrochloride capsules — Anlotinib Hydrochloride is a capsule in the form of 8 mg,10 mg, and 12 mg, orally, once daily, 2 weeks on/1 week off.

SUMMARY:
This is An Open, Single Arm, Multicenter, Exploratory Phase II study, to evaluate the efficacy and safety of TQB2450 Plus anlotinib as adjuvant therapy in hepatocellular carcinoma(HCC) patients at high risk of recurrence after resection. The patients who are confirmed by Histology or cytology as HCC with high-risk recurrence after R0 liver resection will be enrolled. 18 cycles adjuvant treatment with TQB2450 Plus anlotinib can improve one-year recurrence free survival (RFS) rate of HCC patients after R0 surgical resection.

DETAILED DESCRIPTION:
TQB-2450 is a humanized mAb of PD-L1 that prevents PD-L1 from binding to PD-1 and B7.1 receptors on the T cell surface, enabling T cells to restore immune activity and thus enhance the immune response. Anlotinib is a novel multi-target tyrosine kinase inhibitor (TKI) for tumor angiogenesis and proliferative signaling.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation and written informed consent; • Age: 18-75 years old; ECOG PS: 0-1; The expected survival is more than 3 months;
* HCC patients underwent R0 liver resection 4~8 weeks before enrolled; the imaging examination confirmed no recurrence and metastasis according to the RECIST1.1;
* The remaining liver volume must account for more than 40% of the standard liver volume (patients with cirrhosis), or more than 30% (patients without cirrhosis);
* Histologically or cytologically diagnosed as HCC, with any of the following high-risk recurrence conditions: a)Multiple tumor nodules( ≥4 nodules); b)Portal vein tumor thrombosis (PVTT): tumor thrombus distal to the second branches of the portal vein (vp1) and tumor thrombus in the second branches of the portal vein (vp2); c) Portal vein tumor thrombus (PVTT): tumor thrombus in a branch of the hepatic vein (vv1) and tumor thrombus in the right, middle, or left hepatic vein trunk or the short hepatic vein (vv2);
* Laboratory inspection met the following criteria: Hemoglobin (Hb) ≥ 90 g/L, Neutrophils (ANC) ≥ 1.5×10^9/L, Platelet count (PLT) ≥ 75×10^9/L, White blood cell count (WBC) ≥ 3×10^9/L, Total bilirubin (TBIL) ≤ 2.0 × normal upper limit (ULN), Aspartate aminotransferase (AST), and alanine aminotransferase (ALT) ≤ 5.0 ×ULN, Serum creatinine (Cr) ≤ 1.5× ULN, Creatinine clearance rate (CCr) ≥ 60ml/min, International Prothrombin Standardization Ratio (INR) ≤ 1.5 or Prothrombin time (PT) extension < 4s, Thyroid-stimulating hormone (TSH) ≤ULN (patients can be enrolled if the FT3 and FT4 levels are normal);
* Liver function status Child-Pugh grade A(5-6) with no hepatoencephalopathy;
* The woman patients of childbearing age who must agree to take contraceptive methods (e.g. intrauterine device, contraceptive pill, or condom) during the research and within another 6 months after it; who are not in the lactation period and examined as negative in blood serum test or urine pregnancy test within 7 days before the research; The man patients who must agree to take contraceptive methods during the research and within another 6 months after it.

Exclusion Criteria:

* HCC with recurrence after the surgical resection until before enrollment;
* A history of liver cancer resection within 6 months before this surgery;
* Extrahepatic metastasis;
* Diagnosed with cholangiocellular carcinoma, mixed cell carcinoma, and fibrolamellar hepatocellular carcinoma;
* Preoperative treatment with VEGF (R) inhibitors (Anlotinib, sorafenib, Lenvatinib, and so on) or immunomodulator such as anti PD-1, PD-L1, anti CTLA-4;
* Tumor thrombus in the first branch of the portal vein(vp3), tumor thrombus extension to the trunk or the opposite side branch of the portal vein(vp4), tumor thrombus to the inferior vena cava(vv3);
* Patients with chronic active HBV or HCV, HBV-DNA>1000IU/ml, HCV-RNA>1000 copy/ml; hepatitis B with hepatitis C infection;
* Other adjuvant therapy after surgery (except antiviral therapy) ;
* Patients with any severe and/or unable to control diseases;
* The presence of unhealed incisions or fracture;
* A history of gastrointestinal bleeding within 6 months before enrollment; abdominal fistula, gastrointestinal perforation, or abdominal abscess within 2 months before enrollment;
* Standardization Ratio (INR) > 1.5 or Time of partial thrombin activation (APTT) >1.5 × ULN or undergoing thrombolysis or anticoagulation therapy;
* Genetic or acquired bleeding and thrombosis tendency, such as hemophilia, coagulopathy, etc; Patients with arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis, and pulmonary embolism.
* History of another malignancy tumor within 5 years or for now (except for local cancer already cured).
* Patients with a history of immunodeficiency(or autoimmune disease), or other acquired congenital immunodeficiency diseases;
* Local hormone therapy within 2 weeks before treatment;
* Ascites of clinical significance (except for less of Ascites which is asymptomatic)
* Received any live attenuated vaccine within 4 weeks of admission or during the study period;
* Patients who are allergic to components of TQB2450 and anlotinib preparations;
* Patients with concomitant diseases which could seriously endanger their own safety or could affect the completion of the study according to investigators' judgment;
* Failure to follow the study protocol for treatment or scheduled follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
1-year Recurrence-free survival (RFS) rate | 1 year after treatment
  1-year RFS rate is defined as the percentage of patients who do not experience tumor recurrence or death from any cause after 1-year treatment. 1-year RFS rate is determined according to the RECIST 1.1.

SECONDARY OUTCOMES:
Adverse events (AE) | 13 months
  An AE refers to any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, but which does not necessarily have a causal relationship with this treatment. Number and classification of participants with treatment-related adverse events as assessed by CTCAE v5.0 were recorded.
1-year Overall survival (OS) rate | 1 year after treatment
  1-year OS rate is defined as the percentage of patients who do not experience death from any cause after 1-year treatment.
Recurrence-free survival (RFS) | 24 months
  From the date of treatment to the date of diagnosis of tumor recurrence or death from any cause as determined by RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial People's Hospital (The First Affiliated Hospital of Hunan Normal University), Changsha, Hunan, China